CLINICAL TRIAL: NCT04884958
Title: A Prospective Cohort Study to Investigate the Transmission and Burden of PVL-MRSA in Households in Sri Lanka
Brief Title: A Study to Investigate the Transmission and Burden of PVL-MRSA in Households in Sri Lanka
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Sheffield (Other)
Collaborators: Rajarata University, Sri Lanka (Other)
Responsible Party: Sponsor
Other Study IDs: 164460
Record Dates: First submitted 2021-03-03; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-03

CONDITIONS: Staphylococcus Aureus
Keywords: Carriage; Household transmission; MRSA
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Superficial swabs taken from the anterior nares and any clinical sites of infection and then processed for bacterial culture.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Index patient: Adults with confirmed clinical infection caused by Staphylococcus aureus, including skin and soft tissue infection or infection of a normally sterile site. These cases will be identified following admission to Anuradhapura General Hospital.
- Household contacts: This cohort are resident in the same household as the index patient (maximum of four).

SUMMARY:
This study will determine the frequency of Staphylococcus aureus carriage in household contacts of individuals with clinical infection due to this pathogen. It will also assess the frequency of transmission events over the following three months. Finally it will aim to identify predisposing characteristics both on a demographic/social level as well virulence characteristics of the identified strains.

DETAILED DESCRIPTION:
This is a prospective cohort study based at Anuradhapura Teaching Hospital (Sri Lanka). Potential index study participants will have clinical infection caused by Staphylococcus aureus and will be identified from hospital microbiology laboratory records within 48 hours of admission. With consent, the investigators will approach up to 4 household members for participation in the carriage study. With their consent, household members will have swabs collected on 2 occasions 3 months apart. All hospitalised patients will receive standard-of-care treatment in accordance with local practice and national guidance. Clinical, demographic and social/lifestyle data will be collected from index patients and households by scheduled interview performed by local investigators. Bacterial isolates from the initial index patient infection, and those identified through household member screening will be assessed for antimicrobial susceptibility, virulence factor repertoire and analysed by whole genome sequencing. While infection with the cc5 MRSA clone has been described in several hospital and hospital-associated settings in South Asia a major unresolved issue is whether transmission and circulation of this clone is occurring in community settings. In this study the investigators will investigate and characterise the household circulation of Staphylococcus aureus strains, exploring differences in bacterial virulence characteristics and host susceptibility factors associated with increased risk of carriage. Understanding these factors and estimating the burden of disease which may be occurring in the community setting will allow more accurate assessment of the risk posed by cc5 PVL-MRSA to similar Low and Middle Income Countries (LMIC) settings and signal potential routes to mitigation through treatment optimisation and disease prevention including infection control or vaccination.

ELIGIBILITY:
Inclusion Criteria (index patient):

* Confirmed clinical infection caused by Staphylococcus aureus infection, including skin and soft tissue infection (SSTI) or infection of a normally sterile site.
* Participant is willing and able to give informed consent for participation in the study.
* Male or Female greater or equal to 18 years old.
* Household is within one day's travel of the Hospital.

Inclusion Criteria (household contact):

* Resident in the same household as index participant.
* Participant is willing and able to give informed consent for participation in the study if greater or equal to 18 years old or the parent/legal guardian if participant is less than 18 years old.
* Likely continued household residence for at least 3 months from initial sample collection.
* Able to comply with study requirements.

Exclusion Criteria (index patient):

- Deemed unsuitable by the responsible clinical team/clinician (e.g. terminal illness).

Exclusion Criteria (household contact):

* Not a resident of the household at the time of the index patient hospital admission.
* Deemed unsuitable by the responsible clinical team/clinician (e.g. terminal illness)
* At least 4 household contacts already enrolled to this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The index patients will have clinical infection due to Staphylococcus aureus identified during admission to Anuradhapura General Hospital.
  The household contacts will be resident in the same household as the index patient so will be part of the local community served by Anuradhapura General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Determine the baseline prevalence of Staphylococcus aureus carriage or infection in household contacts of hospital inpatients diagnosed with clinical infection due to Staphylococcus aureus. | First household visit and swabbing of household contacts will be as soon as possible after recruitment of the index case.
  Index cases will be identified by screening laboratory reports for samples obtained within 72 hours of hospital admission and where Staphylococcus aureus has been isolated from a skin or soft tissue infection or a normally sterile site and there is a clinical diagnosis of infection at that site. Up to 4 household contacts of this index case will be approached to participate in the study and will have bacterial swabs of the anterior nares and any incidental sites of infection at an initial assessment (as soon after identification and recruitment as possible). The swabs will be inoculated on to blood agar and MacConkey agar. Staphylococcus aureus will be identified by colonial morphology, Gram stain, catalase test and coagulase test. Methicillin resistant Staphylococcus aureus will be detected by disc diffusion method using a cefoxitin disc as per the CLSI protocol.

SECONDARY OUTCOMES:
Measure the frequency of Staphylococcus aureus transmission events within households over a three month period. | First visit and swabbing of the index and household contacts will be as soon as possible after recruitment of the index case. Both the index and household contacts will have a second visit 3 months later (window 2-4 months).
  Proportion of household individuals carrying same/similar strains, as determined by similarity in antimicrobial susceptibility profile and genotypic homology. This will be assessed over a three month time period to detect possible household transmission in contacts who are initially not detected as carriers.
Characterise predisposing clinical, demographic or social characteristic differences of individuals/households with evidence of household transmission over a three month period by interview and completion of a proforma. | The baseline interviews will occur as soon as possible after the index patient is recruited and the second interview will occur three months later (window 2-4 months).
  After consent is obtained, study investigators will visit the dwellings to assess up to 4 household contacts. A baseline interview using a proforma will be conducted to investigate each individual and their shared dwellings. This will include identification of: dwelling location, type of dwelling, number of other inhabitants, pet/animal ownership, occupations, duration of residence, recent illness/hospitalisations, recent courses of antimicrobial treatment. This will be repeated at the follow up visit to ensure there have not been any change in circumstances.
Describe virulence characteristics of strains causing a) (invasive) infection and b) higher number of household transmission events | Data analysis will occur throughout and beyond the study recruitment period, expected to take a minimum of 6 months.
  Analysis of whole genome sequencing and antimicrobial virulence data from isolates that are more associated with infection (in the index and household contacts) and where a high frequency of household transmission has been observed.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Darton, Principal Investigator — University of Sheffield

IPD SHARING:
Plan to Share IPD: Undecided